CLINICAL TRIAL: NCT03805269
Title: Analgesic Efficacy of Ultrasound Guided Transversus Abdominis Plane(TAP) Block Versus Local Anesthetic Infiltration in Adult Patients Undergoing Single Incision Laparoscopic Gastrectomy: A Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane(TAP) Block Versus Local Anesthetic Infiltration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, asociative professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SNUBHTAP
Record Dates: First submitted 2019-01-12; First posted 2019-01-15 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAP block (Experimental): USG guided TAP block
  Interventions: Drug: TAP block
- wound infiltration (Active Comparator): local anesthetics infiltration at surgical incision site
  Interventions: Drug: wound infiltration

INTERVENTIONS:
Drug: TAP block — TAP block: local anesthetics infiltration at trans abdominis plane
  Other Names: TAP
  Arms: TAP block
Drug: wound infiltration — wound infiltration: local anesthetics infiltration at surgical incision
  Other Names: Wound
  Arms: wound infiltration

SUMMARY:
There have been some studies to compared trans abdominis plane(TAP) block with wound infiltration of local anesthetics in multiport laparoscopic surgery, but there have been no studies in single incision laparoscopic gastrectomy.

The purpose of this study was to compare the effect of ultrasonography-guided transverse nerve block and localized anesthesia infiltration in patients with single incision laparoscopic gastrectomy.

DETAILED DESCRIPTION:
Patients were randomly divided into group N(ultrasonography-guided TAP) block and group W( before surgery local anesthetic infiltration at the incision site). We compared the opioid usage, postoperative 6, 24, and 48 hours pain, presence of vomiting, and duration of hospitalization during the operation.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II
* Age: >18

Exclusion Criteria:

* patients of severe kidney & liver dysfunction
* allergy of local anesthetics

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
post operative pain score | 4 hours after end of surgery
  100 mm scale of visual analogue scale

SECONDARY OUTCOMES:
post operative opioid consumption | 4 hours after end of surgery
  total amount of opioid

CONTACTS AND LOCATIONS:
Overall Officials: Jung-hi Ryu, Dr., Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Universuty, Bundang Hospital, Seongnam-si, Gyonggido, South Korea